CLINICAL TRIAL: NCT03716986
Title: Multimodal Imaging of Hypoxia in Gliomas
Acronym: GLIOXYMAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-009
Record Dates: First submitted 2018-10-12; First posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Glioma
Keywords: MRI; Hypoxia; O2 saturation; FMISO PET; Glioma
MeSH Terms: conditions — Glioma; Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SatO2 (Other)
  Interventions: Diagnostic Test: MRI Oxygen Saturation Map

INTERVENTIONS:
Diagnostic Test: MRI Oxygen Saturation Map — Calculation of the oxygen saturation map of gliomas cases

SUMMARY:
The imaging of cerebral oxygenation is an extremely important tool in understanding the pathophysiology of the tumor and for adaptation of therapies according to hypoxia. Currently, imaging of cerebral oxygenation is mainly performed by the use of Positron Emission Tomography (PET). Thus, the investigators have been able to show that the FMISO radiotracer can reveal tumor hypoxia (HypOnco study, promotor: Caen University Hospital, main investigator: J.S. Guillamo). After injection of the radiotracer, increased uptake is observed in the regions for which the tissue oxygen pressure is less than 10 mmHg (the healthy brain with a tissue oxygen pressure (ptO2) ≈ 40mmHg).

Although PET is a reference methodology, it is not widely practiced mainly because of radioactive sources. Magnetic Resonance Imaging (MRI) would bypass the previously mentioned PET limitations. The investigators have recently shown that a measure of local oxygen saturation could be obtained by MRI.

This methodology has also been implemented at a clinical scale on lower field MRI magnets, but its formal validation in a clinical situation remains to be demonstrated with respect to FMISO.

The major advantage of this methodology is that MRI is already performed in routine practice for patients. Measuring tissue oxygenation with MRI (SatO2-MRI) would not add additional examination for the patient. In addition, MRI is a non-ionizing methodology with a very good spatial resolution compared to PET, this should help to better understand intratumoral heterogeneity. Similarly, in preclinical studies, the investigators have shown in a context of mild hypoxia that SatO2-MRI may be more sensitive than PET.

The investigators propose a study to compare in patients with glial tumors, images obtained by 3 Tesla MRI of SatO2-MRI to the hypoxia maps obtained by FMISO PET. These imaging studies will be confronted with studies carried out in immunohistochemistry on biopsies / resection allowing to reveal and to quantify by image analysis the expression of the factors induced by hypoxia (HIF1, HIF2).

This study should include 20 patients with glioma (15 high-grade patients and 5 low-grade patients) in pre-surgery. The aim is to show that SatO2-MRI is a relevant methodology (in terms of sensitivity, specificity) for assessing intratumoral oxygenation in a context of brain tumors. This fits perfectly into an era of personalized medicine where functional imaging finds its meaning.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (> 18 years-old)
* Patient with a diffuse glioma (astrocytoma or oligodendroglioma or glioblastoma)
* Karnofsky index ≥ 70%
* Patient able to understand and sign the consent or accompanied by a trusted person who can do so
* Normal blood test with results: neutrophil ≥ 1500 cells / μl, platelets ≥ 100,000 μl, serum glutamic-oxaloacetic transaminase (SGOT) ≤ 2.5 x upper normal limit (UNL), creatine ≤ 1.5 x UNL
* Patient affiliated to a social security

Exclusion Criteria:

- Patient with contraindications to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
MRI tissue oxygenation map (SatO2-MRI) validation | 7 days
  Validation of SatO2-MRI as a reliable imaging method to detect hypoxic regions, in comparison with FMISO PET. This will mainly be done by measuring spatial correlation of hypoxic regions obtained by the two imaging modalities.

SECONDARY OUTCOMES:
Comparison with pathologic studies | 7 to 90 days
  To correlate imaging biomarkers with more conventional approaches on tissue slices (immunohistochemistry HIF1 / HIF2 / CD34)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Caen, Caen, France